CLINICAL TRIAL: NCT04510415
Title: A Single-arm, Open-label, Phase 1b Study Evaluating the Efficacy and Safety of Olmutinib 600 mg QD in Patients With T790M-positive NSCLC After Treatment With an EGFR-TKI
Brief Title: Olmutinib 600 mg QD in Patients With T790M-positive NSCLC After Treatment With an EGFR-TKI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study termination by the Sponsor
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMSI-103
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — olmutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olmutinib 600mg (Experimental): HM61713 600 mg (1 x 400 mg + 1 x 200 mg tablets) once daily (QD)
  Interventions: Drug: Olmutinib

INTERVENTIONS:
Drug: Olmutinib — 600 mg QD continuously in 21-day cycles until disease progression determined by investigator assessment per RECIST version 1.1, and as long as, in the investigator"s opinion, they are benefiting from study treatment and they do not meet any of treatment discontinuation criteria.
  Other Names: HM61713

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of olmutinib 600 mg QD in patients with T790M-positive non-small cell lung cancer (NSCLC) after treatment with an epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI).

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase 1b study to evaluate the efficacy and safety of oral single agent olmutinib administered to patients with T790M-positive NSCLC after treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before any study-specific procedures (including special Screening tests) are performed.
* At least 20 years of age at the time of signing informed consent.
* Cytologically or histologically confirmed adenocarcinoma of locally advanced or metastatic NSCLC which is not amenable to curative surgery or radiotherapy.
* Radiologically confirmed disease progression after at least one line of treatment with an EGFR-TKI with or without at least one line of chemotherapy.
* At least one documented EGFR mutation which is known to be related with susceptibility to EGFR-TKIs (including G719X, exon 19 deletion, L858R, and L861Q).
* World Health Organization (WHO) performance score of 0 to 1 with life expectancy of at least 3 months.
* Centrally confirmed T790M mutation positive tumor status from a tumor sample taken after confirmation of disease progression on the most recent anticancer treatment regimen.
* At least one lesion (excluding the brain), not previously irradiated that can be accurately measured per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Females of child-bearing potential (not surgically sterilized and between menarche and one-year post-menopause) must agree to use adequate contraception (one of the following listed below) during the study (both men and women as appropriate) and for 3 months after the last dose of study drug.
* Male patients should be documented to be sterile or agree to use barrier contraception i.e. condoms.
* Recovery to ≤ Grade 1 or baseline of any toxicities due to prior treatments, except for stable sensory neuropathy ≤ Grade 2 and alopecia.

Exclusion Criteria:

* Known history of hypersensitivity to active or inactive excipients of HM61713 or drugs with a similar chemical structure of HM61713
* Previous treatment with anticancer therapies, EGFR-TKI (including erlotinib, gefitinib, and afatinib) within 8 days or 5-fold half-life, whichever is the longer, of the first administration of study drug.
* Any non-study related significant surgical procedures within the past 28 days prior to the first administration of study drug
* Spinal cord compression, leptomeningeal carcinomatosis or active symptomatic brain metastases
* History of any other malignancy
* Clinically significant uncontrolled condition(s)
* Active or chronic pancreatitis
* Anyone with cardiac abnormalities or history
* Presence or history of interstitial lung disease (ILD), drug-induced ILD, or presence of radiation pneumonitis.
* Pregnant or breast feeding.
* In the opinion of the investigator, the patient is an unsuitable candidate to receive HM61713.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  Defined as a best overall confirmed response of either CR or PR according to the RECIST version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | 24 months
  Defined as the proportion of patients with a documented CR, PR, and SD during the treatment cycles according to the RECIST version 1.1
Duration of overall tumor response (DR) | 24 months
  Defined as the interval between the date of the first observation of tumor response (CR or PR) and the date of disease progression or death
Progression-free survival (PFS) | 24 months
  Defined as the time from first administration of study drug to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first
Time to progression (TTP) | 24 months
  Defined as the time from first administration of study drug to determination of tumor progression by RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Pharmaceuticals, Study Director — Hanmi Pharmaceuticals
Locations (8):
- South Korea (8):
  - National Cancer Center, Gyeonggi-do
  - The Catholic Univ. of Korea Bucheon St.Mary's Hospital, Gyeonggi-do
  - The Catholic Univ. of Korea St.Vincent's Hospital, Gyeonggi-do
  - The Catholic Univ. of Korea Uijeongbu St.Mary's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - The Catholic Univ. of Korea Incheon St.Mary's Hospital, Incheon
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St.Mary's Hospital, Seoul